CLINICAL TRIAL: NCT05743894
Title: Renal Nerve Simulation Guided Renal Sympathetic Denervation With Siymplicity Spyral Radiofrequency Catheter for Resistant Hypertension: a Feasibility Study.
Brief Title: RDN Fesibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Gormin Tan, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 2022.391
Record Dates: First submitted 2023-02-02; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Hypertension, Renal
Keywords: Renal Sympathetic Denervation; Symplicity Spyral Radiofrequency Catheter; resistant hypertension
MeSH Terms: conditions — Hypertension, Renal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Symplicity Spyral RENAL DENERVATION (RDN) SYSTEMTM Livewire™ Reflexion™ Catheter — Renal sympathetic denervation (RDN) was considered an effective alternative for patients whose blood pressure (BP) is not optimally controlled. The RDN works mainly by selectively ablating the sympathetic fibres around the renal arteries and damping the sympathetic overdrive. Blood pressure response by renal nerve stimulation (RNS) during the RDN procedure using the previous generation of the Symplicity Flex catheter have been reported to be potential parameter to assess the intra-procedure efficacy and predict the BP response 6 months after RDN

SUMMARY:
Renal sympathetic denervation (RDN) was considered an effective alternative for patients whose blood pressure (BP) is not optimally controlled. The RDN works mainly by selectively disabling the nerves around the renal arteries and reducing blood pressure increase. However, despite the early success showed in the SYMPLICITY HTN-2 trial, the SYMPLICITY HTN-3 trial failed to demonstrate a significant BP reduction when compared to sham-control. incomplete disabling might result in inadequate denervation and were cited as some of the contributors to the nil result in the SYMPLICITY HTN-3 . The new generation of the Symplicity Spyral catheter aims to address some of these issues by altering the configuration of the catheter to allow better apposition to the renal arterial wall and increasing the numbers of electrodes to faciiitate more thorough ablations. However, the adequacy of sympathetic denervation with this new catheter can not be easily assessed at the time of the procedure as there is no simple physiological or biochemical feedbacks that can be monitored during the procedure. Blood pressure response by renal nerve simulation (RNS) during RDN procedure using the previous generation of the Symplicity Flex catheter have been reported to be potential parameter to assess the efficacy during the procedure and predict the BP response 6 months after RDN. The feasibility of RNS guided RDN procedure using the new generation of Symplicity Spyral catheter has not been reported. We therefore aim to explore the feasibility of RNS guided RDN with Symplicity Spyral Radiofrequency Catheter in patient with resistant hypertension.

DETAILED DESCRIPTION:
Renal sympathetic denervation (RDN) was considered an effective alternative for patients whose blood pressure (BP) is not optimally controlled. The RDN works mainly by selectively disabling the nerves around the renal arteries and reducing blood pressure increase. However, despite the early success showed in the SYMPLICITY HTN-2 trial, the SYMPLICITY HTN-3 trial failed to demonstrate a significant BP reduction when compared to sham-control. incomplete disabling might result in inadequate denervation and were cited as some of the contributors to the nil result in the SYMPLICITY HTN-3 . The new generation of the Symplicity Spyral catheter aims to address some of these issues by altering the configuration of the catheter to allow better apposition to the renal arterial wall and increasing the numbers of electrodes to faciiitate more thorough ablations. However, the adequacy of sympathetic denervation with this new catheter can not be easily assessed at the time of the procedure as there is no simple physiological or biochemical feedbacks that can be monitored during the procedure. Blood pressure response by renal nerve simulation (RNS) during RDN procedure using the previous generation of the Symplicity Flex catheter have been reported to be potential parameter to assess the efficacy during the procedure and predict the BP response 6 months after RDN. The feasibility of RNS guided RDN procedure using the new generation of Symplicity Spyral catheter has not been reported. We therefore aim to explore the feasibility of RNS guided RDN with Symplicity Spyral Radiofrequency Catheter in patient with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. With resistant hypertension as defined by systolic BP over 140 mmHg on 24 hours ambulatory blood pressure measurement (ABPM)
3. Already on a stable dose of at least 3 anti-hypertensive drugs of different classes for 3 months.
4. subject is recruited for Transcatheter Renal Denervation

Exclusion Criteria:

1. Individual has undergone prior renal denervation.
2. Presence of renal artery stenosis >50%.
3. Main renal artery diameter <3mm and larger than 8mm by visual assessment on angiography.
4. Previous renal stenting.
5. Subject with Estimated GFR <30ml/min/1.73m2 as calculated using the MDRD formula.
6. Subject with renal transplant, single kidney, active nephritis or polycystic kidney disease.
7. Subject with known pheochromocytoma, Cushing's Syndrome (hypercortisolism), primary hyperaldosteronism, coarctation of the aorta, untreated hyperthyroidism, untreated hypothyroidism, or primary hyperparathyroidism.
8. Subject with unstable cardiac conditions such as myocardial infarction, unstable angina, malignant arrythmia, pulmonary embolism, significant valvular condition awaiting surgery or recent cerebrovascular accident within 3 months of recruitment.
9. Subject who is pregnant or planning for pregnancy during the study duration.
10. Subject who is enrolled in another device study for renal sympathetic denervation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a feasibility study, small sample size serves as a proof of concept
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
the difference of RNS BP response before and after RDN | 24-hrs

SECONDARY OUTCOMES:
the changes in 24-hour ABPM after RDN | 6 months
the change in office BP measurement; | 6 months
the change in the number and dosage of anti-hypertensives | 6 months
the change in renal function as measured by estimated GFR | 6 months
the change in renal function as measured by ratio urine albumin-creatinine | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tam GM, Yan BP, Shetty SV, Lam YY. Transcatheter renal artery sympathetic denervation for resistant hypertension: an old paradigm revisited. Int J Cardiol. 2013 Apr 15;164(3):277-81. doi: 10.1016/j.ijcard.2012.01.048. Epub 2012 Feb 14. PMID 22336259
- [Result] Schmieder RE, Mahfoud F, Mancia G, Azizi M, Bohm M, Dimitriadis K, Kario K, Kroon AA, D Lobo M, Ott C, Pathak A, Persu A, Scalise F, Schlaich M, Kreutz R, Tsioufis C; members of the ESH Working Group on Device-Based Treatment of Hypertension. European Society of Hypertension position paper on renal denervation 2021. J Hypertens. 2021 Sep 1;39(9):1733-1741. doi: 10.1097/HJH.0000000000002933. PMID 34261957
- [Result] Weber MA, Mahfoud F, Schmieder RE, Kandzari DE, Tsioufis KP, Townsend RR, Kario K, Bohm M, Sharp ASP, Davies JE, Osborn JW, Fink GD, Euler DE, Cohen DL, Schlaich MP, Esler MD. Renal Denervation for Treating Hypertension: Current Scientific and Clinical Evidence. JACC Cardiovasc Interv. 2019 Jun 24;12(12):1095-1105. doi: 10.1016/j.jcin.2019.02.050. PMID 31221299
- [Result] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Result] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Result] Kandzari DE, Bhatt DL, Brar S, Devireddy CM, Esler M, Fahy M, Flack JM, Katzen BT, Lea J, Lee DP, Leon MB, Ma A, Massaro J, Mauri L, Oparil S, O'Neill WW, Patel MR, Rocha-Singh K, Sobotka PA, Svetkey L, Townsend RR, Bakris GL. Predictors of blood pressure response in the SYMPLICITY HTN-3 trial. Eur Heart J. 2015 Jan 21;36(4):219-27. doi: 10.1093/eurheartj/ehu441. Epub 2014 Nov 16. PMID 25400162
- [Result] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944
- [Result] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589